CLINICAL TRIAL: NCT01928173
Title: Self-Help Video for Insomnia in College Students
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of participants
Sponsor: University of Alabama, Tuscaloosa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-OR-052-ME
Record Dates: First submitted 2013-07-12; First posted 2013-08-23 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2013-08

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: Sleep Initiation and Maintenance Disorders; Cognitive Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abbreviated cognitive behavioral therapy (Active Comparator): Arm 1 is a multi-component package including sleep hygiene, stimulus control, cognitive therapy, and passive relaxation.
  Interventions: Behavioral: Abbreviated cognitive behavioral therapy
- Sleep education/sleep hygiene (Active Comparator): Arm 2 consists of education about sleep and fatigue as well as sleep hygiene recommendations (e.g., avoiding nicotine and caffeine late in the day).
  Interventions: Behavioral: Sleep education/sleep hygiene

INTERVENTIONS:
Behavioral: Abbreviated cognitive behavioral therapy — see arm description
  Arms: Abbreviated cognitive behavioral therapy
Behavioral: Sleep education/sleep hygiene — see arm description
  Arms: Sleep education/sleep hygiene

SUMMARY:
The purpose of this study is to test the effectiveness of a 1-session abbreviated cognitive-behavior therapy for insomnia among college students. The investigators will examine the following hypotheses in the present study: 1) Viewing the treatment video will produce an increment in sleep knowledge relative to baseline and minimum treatment control; and 2) Viewing the treatment video will result in improved sleep relative to baseline and minimum treatment control.

Students who self-identify as having insomnia will be recruited from the University of Alabama's Psychology subject pool. Students who enroll in the study will receive a link to the demographic and screening questionnaire. Individuals who have a history of other sleep disorders or who currently present with symptoms strongly suggestive of sleep disorders, such as obstructive sleep apnea or narcolepsy will be excluded. Individuals who are shift-workers and those with a history of severe mental illness will also be excluded.

Participants who meet criteria for this study will then be directed to complete a measure of sleep knowledge. Once they have completed the measure of sleep knowledge, they will be directed to complete the Consensus Sleep Diary (CSD) for 14 days as soon as possible after awakening in the morning. During the second week of completing the CSD, participants will be directed to complete the Insomnia Severity Index and the Patient-Reported Outcomes Measurement Information System Sleep Disturbance and Sleep-Related Impairments Short Forms on the last day they complete a CSD.

Participants will be randomized to a treatment group or a minimum treatment control group upon completion of these baseline measures. Those in the treatment group will be emailed the following components of the insomnia treatment: a link to the treatment video, an mp3 file with a relaxation recording, and a pdf file of a brochure reviewing the information presented in the treatment video. Participants will be asked to view the treatment video and begin practicing the relaxation technique presented in the mp3 file as soon as possible. Participants in the minimum treatment control group will receive a link to a sleep education video.

Two weeks after participants have viewed the videos, they will be asked to complete post-treatment measures in the same sequence as they did at baseline. One month after the post-treatment measures have been completed, both groups will be asked to complete the same measures again for follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Must be a student at The University of Alabama
* Must be 18-24 years old
* Must have a complaint of insomnia

Exclusion Criteria:

* history of sleep disorder other than insomnia
* symptoms strongly suggestive of sleep disorders other than insomnia
* shift-work
* history of severe mental illness (e.g., psychotic disorders, bipolar disorder, severe depression, or personality disorders)

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Consensus Sleep Diary | Change in sleep diary variables at post-treatment (from baseline to 4 weeks after baseline)
Consensus Sleep Diary | Change in sleep diary variables at 1-month follow-up (post-treatment and 1-month follow-up)

SECONDARY OUTCOMES:
Insomnia Severity Index | Change in score at post-treatment (from baseline to 4 weeks after baseline)
Measure of Sleep Knowledge | Change in number of correct responses at post-treatment (from baseline to 4 weeks after baseline)
  An 8-item true/false questionnaire that assesses participants' knowledge about sleep and cognitive behavioral therapy for insomnia treatment (stimulus control, sleep hygiene, relaxation, and cognitive therapy). A participant's score on this measure is the number of correct responses.
Patient-Reported Outcomes Measurement Information System Sleep Disturbance and Sleep-Related Impairments Short Forms | Change in sleep disturbance and daytime impairments at post-treatment (from baseline to 4 weeks after baseline)
Insomnia Severity Index | Change in score at 1-month follow-up (post-treatment and 1-month follow-up)
Measure of Sleep Knowledge | Change in sleep knowledge at 1-month follow-up (post-treatment and 1-month follow-up)
  An 8-item true/false questionnaire that assesses participants' knowledge about sleep and cognitive behavioral therapy for insomnia treatment (stimulus control, sleep hygiene, relaxation, and cognitive therapy). A participant's score on this measure is the number of correct responses.
Patient-Reported Outcomes Measurement Information System Sleep Disturbance and Sleep-Related Impairments Short Forms | Change in sleep disturbance and daytime impairments at 1-month follow-up (post-treatment and 1-month follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Lichstein, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The University of Alabama, Tuscaloosa, Alabama, United States

REFERENCES:
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Bixler EO, Kales A, Soldatos CR, Kales JD, Healey S. Prevalence of sleep disorders in the Los Angeles metropolitan area. Am J Psychiatry. 1979 Oct;136(10):1257-62. doi: 10.1176/ajp.136.10.1257. PMID 314756
- [Background] Bootzin, R.R., & Epstein, D.R. (2000). Stimulus control instructions. In K.L. Lichstein & C.M. Morin (Eds.), Treatment of late-life insomnia (pp 167-184). Thousand Oaks, CA: Sage.
- [Background] Carney CE, Buysse DJ, Ancoli-Israel S, Edinger JD, Krystal AD, Lichstein KL, Morin CM. The consensus sleep diary: standardizing prospective sleep self-monitoring. Sleep. 2012 Feb 1;35(2):287-302. doi: 10.5665/sleep.1642. PMID 22294820
- [Background] Gustafson R. Treating insomnia with a self-administered muscle relaxation training program: a follow-up. Psychol Rep. 1992 Feb;70(1):124-6. doi: 10.2466/pr0.1992.70.1.124. PMID 1565709
- [Background] Kales JD, Kales A, Bixler EO, Soldatos CR, Cadieux RJ, Kashurba GJ, Vela-Bueno A. Biopsychobehavioral correlates of insomnia, V: Clinical characteristics and behavioral correlates. Am J Psychiatry. 1984 Nov;141(11):1371-6. doi: 10.1176/ajp.141.11.1371. PMID 6496780
- [Background] Morin, C. M. (1993). Insomnia: Psychological assessment and management. New York-London: The Guilford Press.
- [Background] Rosen GM. Self-help treatment books and the commercialization of psychotherapy. Am Psychol. 1987 Jan;42(1):46-51. doi: 10.1037//0003-066x.42.1.46. No abstract available. PMID 3565914
- [Background] Rybarczyk B, Lopez M, Schelble K, Stepanski E. Home-based video CBT for comorbid geriatric insomnia: a pilot study using secondary data analyses. Behav Sleep Med. 2005;3(3):158-75. doi: 10.1207/s15402010bsm0303_4. PMID 15984917
- [Background] Taylor DJ, Gardner CE, Bramoweth AD, Williams JM, Roane BM, Grieser EA, Tatum JI. Insomnia and mental health in college students. Behav Sleep Med. 2011;9(2):107-16. doi: 10.1080/15402002.2011.557992. PMID 21491233